CLINICAL TRIAL: NCT00629044
Title: Etude du Polymorphysme génétique de la cholestérol 24S Hydroxylase et Des Teneurs en 24S hydroxycholestérol Chez Des Patients Atteints de Glaucome ou de dégénérescence Maculaire liée à l'âge.
Brief Title: Genetic Polymorphysm of Cholesterol 24 S Hydroxylase in Patients With Glaucoma and AMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Professor Catherine Creuzot-Garcher, CHU Dijon
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: PHRC IR 2006
Record Dates: First submitted 2008-02-25; First posted 2008-03-05 (Estimated); Last update posted 2011-03-28 (Estimated); Status verified 2009-08

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- G (Active Comparator)
  Interventions: Biological: Assessing the blood level of cholesterol 24 S Hydroxylase
- AMD (Active Comparator)
  Interventions: Biological: Assessing the blood level of cholesterol 24 S hydroxylase
- Healthy subjects (Active Comparator)
  Interventions: Biological: assessing the blood level of cholesterol 24 S hydroxylase

INTERVENTIONS:
Biological: Assessing the blood level of cholesterol 24 S Hydroxylase — Comparison of venous blood level of Cholesterol 24 S hydroxylase and 24 hydroxycholesterol in patients with Glaucoma and AMD and in healthy subjects.
  Arms: G
Biological: Assessing the blood level of cholesterol 24 S hydroxylase — Comparison of venous blood level of cholesterol 24 S hydroxylase and 24 hydroxycholesterol in patients with Glaucoma, AMD end in healthy subjects
  Arms: AMD
Biological: assessing the blood level of cholesterol 24 S hydroxylase — Comparison of venous blood level of cholesterol 24 S hydroxylase and 24 hydroxycholesterol in patients with glaucoma, AMD and in healthy subjects
  Arms: Healthy subjects

SUMMARY:
The aim of this study is to assess the implicitement of the cholesterol 24 S hydroxylase gene and the 24 S hydroxycholesterol in glaucoma and in age related macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Glaucoma
* Patient with AMD
* Healthy patient

Exclusion Criteria:

* All patients who use any treatment in order to maintain in normal value their blood cholesterol

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2007-11; Primary Completion 2009-11 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To know if cholesterol 24 S hydroxylase and 24 hydroxycholesterol are involve in Glaucoma and AMD | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Creuzot-Gracher, MD, PhD, Principal Investigator — CHU Dijon
Locations (1):
- Ophthalmology Unit CHU Dijon, Dijon, Burgundy, France

REFERENCES:
- [Background] Joffre C, Souchier M, Gregoire S, Viau S, Bretillon L, Acar N, Bron AM, Creuzot-Garcher C. Differences in meibomian fatty acid composition in patients with meibomian gland dysfunction and aqueous-deficient dry eye. Br J Ophthalmol. 2008 Jan;92(1):116-9. doi: 10.1136/bjo.2007.126144. PMID 18156378